CLINICAL TRIAL: NCT03319628
Title: A Phase 1b/2, First-in-Human, Dose Escalation and Expansion Study of XMT-1536 In Patients With Solid Tumors Likely to Express NaPi2b
Brief Title: First-in-Human Study of XMT-1536 in Cancers Likely to Express NaPi2b
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mersana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XMT-1536-1
Record Dates: First submitted 2017-10-17; First posted 2017-10-24 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-09

CONDITIONS: Platinum Resistant Ovarian Cancer; Non Small Cell Lung Cancer Metastatic

STUDY DESIGN:
Intervention Model Description: Open-label, dose escalation to reach MTD. The MTD will be confirmed in parallel cohorts: patients with platinum-resistant ovarian cancer; patients with non-squamous NSCLC, adenocarcinoma subtype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Escalation (Experimental): XMT-1536 (upifitamab rilsodotin) treatment is administered in groups of patients who will receive doses that increase over time.
  This cohort is closed to enrollment.
  Interventions: Drug: upifitamab rilsodotin
- Dose Expansion - Ovarian Cancer (Experimental): Once the maximum tolerated dose or recommended Phase 2 dose is achieved in dose escalation, new groups of patients will receive XMT-1536 (upifitamab rilsodotin) at this fixed-dose.
  This cohort is closed to enrollment.
  Interventions: Drug: upifitamab rilsodotin
- Dose Expansion - NSCLC adenocarcinoma (Experimental): Once the maximum tolerated dose or recommended Phase 2 dose is achieved in dose escalation, new groups of patients will receive XMT-1536 (upifitamab rilsodotin) at this fixed-dose.
  This cohort is closed to enrollment.
  Interventions: Drug: upifitamab rilsodotin
- Pivotal Cohort (UPLIFT) (Experimental): Patients with platinum-resistant ovarian cancer will receive XMT-1536 (upifitamab rilsodotin) to further confirm the efficacy.
  This cohort is closed to enrollment.
  Interventions: Drug: upifitamab rilsodotin
- QTc Sub-Study (Experimental): For sites participating in the sub-study, patients with platinum -resistant ovarian cancer will have the option to enroll in this sub-study to evaluate potential changes in the QTc interval following administration of XMT-1536.
  This cohort is closed to enrollment.
  Interventions: Drug: upifitamab rilsodotin

INTERVENTIONS:
Drug: upifitamab rilsodotin — XMT-1536 will be administered once every 28 days until disease progression, unacceptable toxicity, or either the patient or study physician determines it is in the best interest of the patient to discontinue participation in the study.
  For sites participating in the sub-study, patients with platinum -resistant ovarian cancer will have the option to enroll in this sub-study to evaluate potential changes in the QTc interval following administration of XMT-1536
  Other Names: XMT-1536; UpRi

SUMMARY:
First-in-human, Phase 1b/2 safety study of the antibody-drug conjugate (ADC) XMT-1536 (upifitamab rilsodotin) administered as an intravenous infusion once every four weeks. Patients with tumor types likely to express NaPi2b were enrolled in dose escalation. Patients with platinum-resistant ovarian cancer and non-small cell lung cancer (adenocarcinoma subtype) were enrolled in the expansion segment of this study. Patients with platinum-resistant, high-grade serous ovarian cancer were enrolled in the UPLIFT segment of this study. In addition to safety assessments, the pharmacokinetics of the drug were assessed along with ADC activity. A QTc sub-study was added for the UPLIFT cohort for a sub-set of sites.

DETAILED DESCRIPTION:
This is a multi-center study of XMT-1536 (upifitamab rilsodotin) in patients with tumors likely to express NaPi2b, focusing on patients with platinum-resistant ovarian cancer and non-small cell lung cancer, adenocarcinoma subtype. XMT-1536 (upifitamab rilsodotin) was administered as an intravenous infusion once every four weeks. The study consisted of three segments: dose escalation (DES), dose expansion (EXP), and the pivotal cohort (UPLIFT). The DES segment studied small groups of patients who received increased doses. A Safety Review Committee was established to review the data from each dose level before moving to the next higher dose. The dose escalation cohort has ended and is no longer enrolling patients. Enrollment into the EXP segment consisted of 2 parallel cohorts of patients to confirm the dose that has been identified in DES and estimate the objective response rate in each patient population. The EXP and UPLIFT cohorts are no longer enrolling patients. All adverse events were graded according to the National Cancer Institute (NCI) Common Terminology Criteria version (CTCAE v5.0). Throughout the study, pharmacokinetics were measured using proprietary assays developed by Mersana. Anti-cancer activity were measured via RECIST.

ELIGIBILITY:
General Inclusion Criteria (for Dose Escalation, Expansion, and UPLIFT):

* ECOG performance status 0 or 1
* Measurable disease as per RECIST, version 1.1
* Resolution of all acute toxic effects of prior therapy or surgical procedures to ≤Grade 1 (except alopecia, stable immune-related toxicity such as hypothyroidism on hormone replacement, adrenal insufficiency on ≤10 mg daily prednisone [or equivalent], chronic Grade 2 peripheral sensory neuropathy after prior taxane therapy).
* Cardiac left ventricular ejection fraction (LVEF) ≥50% or ≥ the institution's lower limit of normal by either Echo or MUGA scan
* Adequate organ function as defined by the following criteria:

  1. Absolute neutrophil count (ANC) ≥1500 cells/mm3
  2. Platelet count ≥100,000/mm3
  3. Hemoglobin ≥9 g/dL
  4. In patients not on anticoagulation therapy: INR, activated partial thromboplastin time (aPTT), and prothrombin time (PT) all within 1.2 times the institution's upper limit of normal (ULN). Patients on anticoagulation therapy are allowed if their relevant laboratory values are within the therapeutic window.
  5. Estimated glomerular filtration rate (GFR) ≥45 mL/min
  6. Total bilirubin ≤ULN
  7. g. Patients with asymptomatic elevations in unconjugated bilirubin due to Gilbert syndrome or stable chronic hemolytic anemia (e.g., hereditary spherocytosis, sickle cell disease, thalassemia intermedia) may be eligible after discussion with the Sponsor Medical Monitor.
* Aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤1.5 times the institutional ULN.
* Albumin ≥3.0 g/dL
* Able to provide informed consent.

General Exclusion Criteria (for Dose Escalation, Expansion, and UPLIFT) :

* Major surgery within 28 days of starting study treatment, systemic anti-cancer therapy within the lesser of 28 days or 5 half-lives of the prior therapy before starting study treatment, or recent radiation therapy with unresolved toxicity or within a time window of potential toxicity.
* Patients with untreated CNS metastases (including new and progressive brain metastases), history of leptomeningeal metastasis or carcinomatous meningitis.
* Current known active infection with HIV, hepatitis B virus, or hepatitis C virus.
* Prior history of liver disease such as liver cirrhosis, hepatic fibrosis
* Current severe, uncontrolled systemic disease (e.g., clinically significant cardiovascular, pulmonary, or metabolic disease) or intercurrent illness that could interfere with per-protocol evaluations.
* Current use of either constant or intermittent supplementary oxygen therapy.
* History of suspected pneumonitis or interstitial lung disease.
* Pregnant or nursing women.
* History of other malignancy within the last 2 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or other malignancy with a similar expected curative outcome.
* Active corneal disease, or history of corneal disease within 12 months prior to enrollment
* Use of strong CYP450 3A inhibitors or inducers that cannot be discontinued while receiving study treatment
* Oxygen saturation on room air <93%

Ovarian Cancer Inclusion Criteria for UPLIFT:

* Histological diagnosis of high grade serous ovarian cancer, which includes fallopian tube, or primary peritoneal cancer, that is metastatic or recurrent.
* Platinum-resistant disease

  1. Patients who have only had 1 line of platinum-based therapy must have received at least 4 cycles of platinum, must have had a response [complete response/remission (CR) or partial response/remission (PR)], and then progressed between 3 months and ≤ 6 months after the date of the last dose of platinum
  2. Patients who have received 2 to 4 lines of prior therapy must have received at least 4 cycles of platinum and then progressed within 6 months after the date of the last dose of platinum
* One to 4 prior lines of systemic therapy for ovarian cancer

  a. Prior treatment with bevacizumab is required for patients with 1 to 2 prior lines of therapy
* Patients must be willing to provide an archival tumor tissue block or slides or if not available, undergo procedure to obtain a new tumor biopsy using a low-risk, medically routine procedure

Ovarian Cancer Exclusion Criteria for UPLIFT:

* Low-grade, clear cell, endometrioid, mucinous, carcinosarcoma, germ-cell, mixed histology, or stromal tumors
* Prior treatment with mirvetuximab soravtansine or another ADC containing an antitubulin payload
* Primary platinum-resistant disease, defined by a lack of response or by progression within 3 months after completing front-line, platinum-containing therapy.
* Participation in DES or EXP segments of this study

Ovarian Cancer Inclusion Criteria for QTc sub-study:

Note: patients must meet all UPLIFT cohort inclusion criteria in order to participate in the QTc sub-study

• Study patient has agreed to remain in the clinic for the additional QTc related study activities on the Day 1 of Cycle 1 and Cycle 3.

Ovarian Cancer Exclusion Criteria for QTc sub-study:

* Use of strong CYP450 3A inducers.
* Uncontrolled cardiac arrhythmias, for example, atrial fibrillation with a ventricular response at rest > 100 beats per minute. left bundle branch block (LBBB)
* Known abnormality of any cardiac valve (either stenosis or regurgitation) that is greater than moderate in severity.
* Subjects not in sinus rhythm at screening with HR >45- <100
* Any ECG abnormality that can interfere with the measurement of the QT interval

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 523 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
DES: Maximum tolerated dose or recommended Phase 2 dose | Up to 36 weeks, from the date of first dose until unacceptable side effects or a dose-limiting toxicity is met
  Evaluate adverse events and concomitant medication use after XMT-1536 (upifitamab rilsodotin) doses
DES and EXP: Safety and Tolerability | First dose up until 30 days after study termination
  Evaluate incidence and severity of adverse events
EXP: Anti-neoplastic effects of XMT-1536 (upifitamab rilsodotin) | Every 6 weeks for up to 36 weeks
  Monitor tumor size
UPLIFT: Investigator-assessed objective response rate (ORR) of XMT-1536 (upifitamab rilsodotin) in the ITT-Higher NaPi2b population | Every 8 weeks until disease progression or up to 24 months
  Confirmed ORR is defined as the proportion of patients who have achieved a confirmed complete response (CR) or partial response (PR) per RECIST v1.1 after the initiation of study treatment.
QTc Sub-study: Evaluation of the concentration response analysis of XMT-1536 versus the change in QTcF values | 60 minutes prior to first dose, up to 26 hours after Cycle 3 dose
  "The concentration-QTcf change from baseline deltaQTcF analysis and analysis of central tendency for deltaQTcF

SECONDARY OUTCOMES:
DES and EXP: Time of maximum observed concentration of XMT-1536 (upifitamab rilsodotin) | Daily for one week after first dose; weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1536 (upifitamab rilsodotin)
DES and EXP: Maximum concentration of XMT-1536 (upifitamab rilsodotin) | Daily for one week after first dose; weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1536 (upifitamab rilsodotin)
DES and EXP: Area under the concentration curve of the last measurable concentration of XMT-1536 (upifitamab rilsodotin) | Daily for one week after first dose; weekly until 28 days after first dose; immediately before and after and 1 week after all subsequent doses
  Determine the pharmacokinetics of XMT-1536 (upifitamab rilsodotin)
DES: Anti-neoplastic effects of XMT-1536 (upifitamab rilsodotin) | Every 6 weeks for up to 36 weeks
  Monitor tumor size
DES and EXP: Anti-drug antibody and neutralizing antibody | Every 6 weeks for up to 36 weeks
  Analyze blood for antibodies to XMT-1536 (upifitamab rilsodotin) and neutralizing antibodies
UPLIFT: Confirmed Investigator-assessed objective response rate of XMT-1536 (upifitamab rilsodotin) regardless of NaPi2b expression | Every 8 weeks until disease progression or up to 24 months
  Assess the confirmed investigator-assessed objective response rate of XMT-1536 (upifitamab rilsodotin) regardless of NaPi2b expression
UPLIFT: Confirmed objective response rate by independent radiology review (IRR) for patients with high NaPi2b and overall | Every 8 weeks until disease progression or up to 24 months
  Assess the confirmed objective response rate by IRR for patients with high NaPi2b (TPS >/=75) and overall
UPLIFT: Duration of objective response (DOR) | 4 weeks after first response and every 8 weeks until disease progression or up to 24 months
  Assess the duration of objective response (DOR) in patients who achieve a response
UPLIFT: Incidence and severity of adverse events | First dose up until 60 days after study termination
  Evaluate incidence and severity of adverse events
QTc Sub-Study: Evaluation of the effect of XMT-1536 on QTcF in patients with platinum-resistant HGSOC by timepoint analysis | 60 minutes prior to first dose, up to 26 hours after Cycle 3 dose
  Con.-QTc evaluation
QTc Sub-Study: Evaluation of the effect of XMT-1536 on the PR-interval (PR), QRS duration (QRS), Heart Rate (HR), and ECG morphology | 60 minutes prior to first dose, up to 26 hours after Cycle 3 dose
  Con.-QTc evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Burger, MD, Study Director — Mersana Therapeutics
Locations (1):
- University of Oklahoma, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No